CLINICAL TRIAL: NCT05906550
Title: Flow Dysfunction of Hemodialysis Vascular Access: a Randomized Controlled Trial on the Effectiveness of Surveillance of Arteriovenous Fistulas and Grafts
Brief Title: Flow Dysfunction of Hemodialysis Vascular Access
Acronym: FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL75845.068.20; NL9165 (Registry Identifier: Netherlands Trial Registry)
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dialysis Access Malfunction; Hemodialysis Access Failure; Hemodialysis Fistula Thrombosis; Vascular Access Malfunction

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial with hybrid parallel-crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The software of the HD03 Hemodialysis Monitor will be adjusted to allow blinded measurements that will be sent to the trial coordinator; patients and health care providers remain unaware of treatment allocation and surveillance findings. Flow measurements will only be used to refer patients for correction of vascular access stenosis in the control group. To maintain blinding, whenever a measurement must be repeated to confirm low flow volumes, another trial participant will randomly be selected for confirmation of vascular access flow volumes after the next measurement. Patients will be censored and randomized anew following an intervention for flow dysfunction, as soon as the indicator for vascular access intervention has been resolved and vascular access function has been restored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients are referred for correction of the underlying stenosis when clinical signs of flow dysfunction are present. These include physical signs, problems during dialysis, or an unexplained, sustained fall in dialysis adequacy.
  Interventions: Diagnostic Test: Vascular access monitoring
- Control group (Active Comparator): Monthly surveillance of vascular access blood flow volume by ultrasound dilution measurements during hemodialysis sessions. Patients will be referred for correction of the underlying stenosis at an access flow volume <500mL/min, or when clinical signs of flow dysfunction are present.
  Interventions: Diagnostic Test: Vascular access monitoring; Diagnostic Test: Vascular access blood flow measurement

INTERVENTIONS:
Diagnostic Test: Vascular access monitoring — Patients are referred for correction of the underlying stenosis when clinical signs of flow dysfunction are present. These include physical signs, problems during dialysis, or an unexplained, sustained fall in dialysis adequacy. Patients will be referred for correction of the underlying stenosis when clinical signs of flow dysfunction are present.
Diagnostic Test: Vascular access blood flow measurement — Monthly surveillance of vascular access blood flow volume by ultrasound dilution measurements during hemodialysis sessions. Patients will be referred for correction of the underlying stenosis at an access flow volume <500mL/min.
  Arms: Control group

SUMMARY:
The FLOW trial evaluates the follow-up of the vascular access for hemodialysis. In current clinical care, vascular access flow volume is periodically assessed to detect and treat asymptomatic stenosis. The FLOW trial will determine whether it is safe to abandon this practice of active surveillance. Vascular access stenosis will then be treated only when clinical problems of flow dysfunction occur during hemodialysis. The investigators expect that the intervention rate and medical costs will be reduced by 40% when correction of vascular access stenosis is triggered by clinically apparent access dysfunction rather than asymptomatic flow reduction.

DETAILED DESCRIPTION:
Study design: Multicenter randomized controlled trial with 375 patients. Patients will be followed up for 2 to 3 years. The trial is powered to detect a reduction in the intervention rate of 0.25 per year between study groups in a superiority analysis (this is associated with cost savings of 1 million euros per year in the Netherlands). Subgroup analyses of arteriovenous fistulas and grafts and of successful and failed interventions will be done.

On 25-02-2025, the sample size was reduced from 417 to 375 patients because updated calculations based on actual event and loss to follow-up rates in the trial population showed sufficient power to detect the prespecified clinically relevant difference.

Study population: Chronic hemodialysis patients with a functioning arteriovenous fistula or graft.

Intervention group: Patients are referred for correction of the underlying stenosis when clinical signs of flow dysfunction are present. These include physical signs, problems during dialysis, or an unexplained, sustained fall in dialysis adequacy.

Control group: Monthly surveillance of vascular access blood flow volume by ultrasound dilution measurements during hemodialysis sessions. Patients will be referred for correction of the underlying stenosis at an access flow volume <500mL/min, or when clinical signs of flow dysfunction are present.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years or older.
2. End-stage renal disease with unlikely recovery of kidney function according to the attending nephrologist.
3. Arteriovenous fistula or arteriovenous graft as hemodialysis vascular access that fulfills both of the following criteria at the time of trial enrollment:

   1. Vascular access flow volume of at least 500mL/min; and
   2. Functional vascular access: the vascular access was cannulated with 2 needles and achieved the prescribed access circuit flow in at least 6 dialysis sessions over the past 30 days. Patients who have single needle hemodialysis for reasons other than vascular access dysfunction (e.g. for nocturnal hemodialysis) but who can be cannulated with 2 needles for flow measurements and fulfill the other requirements for a functional vascular access can be enrolled as well.
4. Planning to remain in one of the participating dialysis centers for at least 1 year.

Exclusion Criteria:

1. Arteriovenous fistulas with multiple venous outflow paths upstream of the cannulation sites, that are not suitable for flow volume measurements using ultrasound dilution (e.g. Gracz fistulas and Ellipsys or WavelinQ endovascular fistulas).
2. Home hemodialysis.
3. Thrombosis of the current vascular access in the past year.
4. Planned access-related intervention.
5. Living donor kidney transplantation, switch to peritoneal dialysis, or switch to home hemodialysis planned within 6 months.
6. Life expectancy of less than 6 months, in the opinion of the attending nephrologist.
7. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Access-related intervention rate | Variable follow-up time of 2-3 years
  The number of interventions required for each patient-year of hemodialysis treatment

SECONDARY OUTCOMES:
Access-related complications per patient-year (1) | Variable follow-up time of 2-3 years
  Clavien-Dindo grade 2 complications (requiring pharmacological treatment)
Access-related complications per patient-year (2) | Variable follow-up time of 2-3 years
  Access-related serious adverse events (Clavien-Dindo grade 4 and 5 complications, and vascular access thrombosis)
All-cause mortality | Variable follow-up time of 2-3 years
  All-cause mortality
Access-related health care costs (1) | Every 3 months for 2-3 years from randomization (variable follow-up time)
  Medical Consumption Questionnaire
Access-related health care costs (2) | Every 3 months for 2-3 years from randomization (variable follow-up time)
  Productivity Cost Questionnaire
Patient-reported outcome measures (1) | Every 3 months for 2-3 years from randomization (variable follow-up time)
  SF-VAQ (Short-Form Vascular Access Questionnaire)
Patient-reported outcome measures (2) | Every 3 months for 2-3 years from randomization (variable follow-up time)
  EQ-5D-5L
Quality of the surveillance program (1) | Variable follow-up time of 2-3 years
  Repeatability and reproducibility of vascular access flow volume measurements
Quality of the surveillance program (2) | Variable follow-up time of 2-3 years
  Diagnostic accuracy of vascular access flow volume measurements to predict clinical signs of flow dysfunction and access thrombosis within 1 month in the intervention group
Quality of the surveillance program (3) | Variable follow-up time of 2-3 years
  The percentage of vascular access balloon angioplasties resulting in technical success (residual stenosis <30%) and clinical success (increase in flow volume to >500mL/min, restoration of vascular access function and resolution of any clinical signs of flow dysfunction)
Quality of the surveillance program (4) | Variable follow-up time of 2-3 years
  Vascular access patency after balloon angioplasty
Primary patency | Variable follow-up time of 2-3 years
  This outcome measure will be registered for explanatory analyses
Assisted primary patency | Variable follow-up time of 2-3 years
  This outcome measure will be registered for explanatory analyses
Secondary patency | Variable follow-up time of 2-3 years
  This outcome measure will be registered for explanatory analyses
The number of hemodialysis sessions with cannulation difficulties | Variable follow-up time of 2-3 years
  This outcome measure will be registered for explanatory analyses

CONTACTS AND LOCATIONS:
Overall Officials: Maarten G Snoeijs, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (13):
- Netherlands (13):
  - Diapriva - Dialyse Centrum Amsterdam, Amsterdam
  - OLVG, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - Medisch Spectrum Twente, Enschede
  - Spaarne Gasthuis, Haarlem
  - Zuyderland Medisch Centrum, Heerlen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht UMC+, Maastricht
  - Bravis Ziekenhuis, Roosendaal
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
The size of the data collection is unknown but includes physical examination forms, Transonic flow measurement curves, angiography videos, and intervention notes.
  The following end products will be made available for further research and verification: data documentation; documentation of the research process, including documentation of all participants; audiovisual material / images; several versions of processed data; raw data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The embargo period will be as long as required for publication of the research findings.
Access Criteria: Interested parties can submit a request for a data set.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT05906550/SAP_000.pdf